CLINICAL TRIAL: NCT03242629
Title: Effects Comparison Between Oral and Enema of Chloral Hydrate in Pediatric Ophthalmic Examination
Brief Title: Comparison Between Oral and Enema of Chloral Hydrate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Haotian Lin, Clinical Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CCPMOH2017-China-6
Record Dates: First submitted 2017-07-30; First posted 2017-08-08 (Actual); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Congenital Cataract
Keywords: pediatric ophthalmic examination; chloral hydrate; Effects Comparison
MeSH Terms: interventions — Chloral Hydrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- oral group (Active Comparator)
  Interventions: Drug: oral chloral hydrate
- enema group (Experimental)
  Interventions: Drug: enema chloral hydrate

INTERVENTIONS:
Drug: oral chloral hydrate — Chloral hydrate syrup was available in a concentration of 100 mg×ml-1.The children assigned to receive 0.8 ml×kg-1 of chloral hydrate (80 mg×kg-1) by oral.
  Arms: oral group
Drug: enema chloral hydrate — Chloral hydrate syrup was available in a concentration of 100 mg×ml-1 at our hospital.The children assigned to receive 0.8 ml×kg-1 of chloral hydrate (80 mg×kg-1) by enema.
  Arms: enema group

SUMMARY:
To compare the clinical sedative effect and safety using 10% chloral hydrate during ophthalmic examinations for oral vs enema group.The patients were randomly divided into two groups (oral group and enema group) using a computer random number generator with a 1:1 allocation (simple randomization, odd number for oral group and even number for enema group).

DETAILED DESCRIPTION:
To compare the clinical sedative effect and safety using 10% chloral hydrate during ophthalmic examinations for oral vs enema group.The patients were randomly divided into two groups (oral group and enema group) using a computer random number generator with a 1:1 allocation (simple randomization, odd number for oral group and even number for enema group).One hundred and twenty children aged from 3 to 36 months (5-15 kg) scheduled to ophthalmic examinations were randomly sedated by oral chloral hydrate(80 mg×kg-1, n = 60) or enema chloral hydrate(80 mg×kg-1, n = 60). The primary endpoint was successful sedation to complete the examinations including slit-lamp photography, tonometry, anterior segment analysis, and refractive error inspection. The secondary endpoints included onset time, duration of examination, recovery time, discharge time, any side effects during examination, and within 48 h after discharge.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with congenital cataract aged from 3 to 36 months weight from 5 to 15 kg with American Society of Anesthesiologists (ASA) physical status 1-2

Exclusion Criteria:

* with gastro-esophageal reflux, nausea and vomiting, apnea in the past 3 months recent pneumonia exacerbation of asthma, bronchitis and upper respiratory tract infection bradycardia, and facial abnormalities, allergy to chloral hydrate, weight <2 or >20 kg .

Ages: 3 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Demography (age, sex, weight， laterality and medical history) | baseline
  The demography of cataract and healthy children were recorded by using a semi-structured questionnaire

SECONDARY OUTCOMES:
Side effect | the following 48 hour after using the drug
  record the following symptom: Vomit after administration、Cough、SpO2 < 95%、SpO2 < 90%、New vomiting、Resume normal activity over 8 hour、Poor appetite、Altered bowel habit
the time of Sleepiness:Onset time (min） | baseline
the time of Sleepiness:Duration of examination (min) | baseline
the time of Sleepiness:Recovery time (min) | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Haotian Lin, M.D,Ph.D, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University